CLINICAL TRIAL: NCT01587794
Title: Topographic Changes of Retinal Layers After Resolution of Acute Retinal
Brief Title: Topographic Changes of Retinal Layers After Resolution of Acute Retinal Detachment
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Se Woong, Kang, M.D., Samsung Medical Center
Other Study IDs: 2011-3-31
Record Dates: First submitted 2012-03-31; First posted 2012-04-30 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: Rhegmatogenous retinal detachment; thickness of retinal layer; outer nuclear layer; photoreceptor layer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- retinal detachment group: Patients who were diagnosed with unilateral rhegmatogenous retinal detachment involving only the superior or inferior half of the retina and who underwent successful scleral buckling procedure or vitrectomy by a single surgeon between January 1, 2008 and April 1, 2010 were included in the study sample.

SUMMARY:
Experimental retinal detachment and reattachment models have demonstrated the recovery process of successfully reattached retina. However, optical coherence tomography analysis of each retinal layers following retinal reattachment has not been investigated This study investigated changes in thickness profiles of retinal layers after resolution of recent-onset rhegmatogenous retinal detachment (RRD) using optical coherence tomography images.

DETAILED DESCRIPTION:
Rhegmatogenous retinal detachment is a sight-threatening condition that occurs when the neurosensory retina separates from the underlying retinal pigment epithelium and fluid accumulates within this potential space.Surgical reattachment of a detached retina is the mainstay of treatment.

Experimental retinal detachment and reattachment models have demonstrated the recovery process of successfully reattached retina, including regrowth and reconfiguration of the photoreceptor inner and/or outer segments,reorganization of photoreceptor-RPE interface,increased synaptic terminals in the outer plexiform layer, inhibition of glial cell proliferation,and recovery of normal distribution of proteins. These microscopic changes are thought to be the reason for visual function recovery following retinal reattachment.

Recent development in spectral domain optical coherence tomography, which provides faster imaging speed and higher resolution, allows more detailed retinal layer evaluation. Previous studies using spectral domain optical coherence tomography have revealed abnormalities of retinal microstructure in reattached retina. However, these studies mainly focused on the photoreceptor layer and/or external limiting membrane, although abnormalities of various retinal layers have been revealed in previous microscopic studies. In addition, qualitative rather than quantitative analysis was performed in most of the studies, and most importantly, all previous studies were observational and comparisons between the affected and normal control regions were not performed.

The current study involves a series of recent-onset primary rhegmatogenous retinal detachment that were managed with surgical retinal reattachment. The investigators quantified the thickness of each retinal layer based on spectral domain optical coherence tomography images and compared the thicknesses of reattached regions and undetached normal regions. The primary purpose of this study was to evaluate the changes in thickness profiles of each retinal layer in reattached retina after acute RRD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who could estimate the time of onset of visual symptom of retinal detachment (sudden decrease in visual acuity or onset of visual field defect) accurately
* Patients who were treated within 2 weeks of symptom onset Exclusion Criteria:

Exclusion Critetia:

* traumatic retinal detachment
* recurred retinal detachment
* less than 6 months of follow-up after surgery
* insufficient cooperation for optical coherence tomography examination
* media opacity that would preclude acquisition of clear optical coherence tomography images
* -6.0 diopters or more of spherical equivalent
* prominent staphyloma
* history of intraocular surgery other than cataract surgery or intraocular lens implantation
* other ocular diseases that may influence the macular microstructure.
* individuals with indistinct intraretinal structure on optical coherence tomography images
* large retinal vessels at the location of thickness measurement, or epiretinal membrane

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed with unilateral RRD involving only the superior or inferior half of the retina and who underwent successful scleral buckling procedure or vitrectomy by a single surgeon between January 1, 2008 and April 1, 2010 were included in the study sample.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Thickness of each retinal layer | At least 6 months after the operation
  SD-OCT scans were performed for all patients enrolled using Spectralis optical coherence tomography. The thickness of each retinal layer was measured manually using the included Heidelberg Eye Explorer software.

REFERENCES:
- [Derived] Kim JH, Park DY, Ha HS, Kang SW. Topographic changes of retinal layers after resolution of acute retinal detachment. Invest Ophthalmol Vis Sci. 2012 Oct 23;53(11):7316-21. doi: 10.1167/iovs.12-10155. PMID 23033395